CLINICAL TRIAL: NCT00847951
Title: 3D Ultrasound for Perfusion in Neonates
Brief Title: Ultrasound for Perfusion in Neonates
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated at this time by investigator. Will create new protocol.
Sponsor: University of Michigan (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Jonathan Rubin, M.D., Principal Investigator, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM00021322
Record Dates: First submitted 2009-02-17; First posted 2009-02-19 (Estimated); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Kidney Perfusion
Keywords: renal; neonates

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Renal perfusion in Neonates (Other): Ultrasound scanning with power Doppler is used to determine the fractional blood volume of the kidneys.
  Interventions: Procedure: 3D Ultrasound Imaging

INTERVENTIONS:
Procedure: 3D Ultrasound Imaging — Ultrasound scanning with power Doppler is used to determine the fractional blood volume of the kidneys in pre-mature and/or very low birth weight babies. This is a measure of perfusion and an indication of how well the kidneys are working.

SUMMARY:
The purpose of this study is to evaluate the effectiveness of renal ultrasound to check kidney perfusion in premature and/or very low birth weight babies.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effectiveness of 3D (3 dimensional)renal ultrasound to check kidney perfusion (to see if the kidney is receiving enough blood flow to function as it should) in premature and/or very low birth weight babies.

ELIGIBILITY:
Inclusion Criteria:

* Very low birth weight babies in ICU in stable condition and/or premature babies in ICU in stable condition

Exclusion Criteria:

* Unstable very low birth weight/premature babies

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2008-10 (Actual); Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
To determine if ultrasound imaging can accurately help physicians determine if the kidneys are being adequately perfused. | 1 year
  Fractional blood volume was determined as a way to measure kidney perfusion. Adequate perfusion indicates that the kidneys are working and might indicate if a baby was responding to a specific treatment or not.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Rubin, MD, Principal Investigator — Univeristy of Michigan Hospital
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No